CLINICAL TRIAL: NCT01553383
Title: Comparison of Nasal Positive End Expiratory Pressure Valve to Dental Device as an Alternative Treatment for OSA
Brief Title: Comparison of Nasal Positive End Expiratory Pressure Valve to Dental Device as an Alternative Treatment for Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, To Kin Wang, Associate consultant, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CREC2012.037
Record Dates: First submitted 2012-03-01; First posted 2012-03-14 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Obstructive Sleep Apnea; Adverse Effects
Keywords: OSA
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dental device (Active Comparator): "Provent" nasal peep valve vs dental device
  Interventions: Device: nasal peep valve "Provent"
- CPAP (Active Comparator): continuous positive airway pressure "CPAP" vs nasap peep valve "Provent"
  Interventions: Device: nasal peep valve "Provent"

INTERVENTIONS:
Device: nasal peep valve "Provent" — application of nasal peep valve vs dental device and cpap

SUMMARY:
Determine the clinical efficacy in terms of Apnea Hypopnea Index (AHI), excessive daytime sleepiness (EDS), nocturnal oxygenation of a nasal Positive end-expiratory pressure (PEEP) valve "Provent" in obstructive sleep apnea. The hypothesis is the efficacy will be better than dental device.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic patients confirmed of OSA by sleep study (PSG according to AASM criteria or validated level 3 portable monitoring devices with AHI > 10/hr)
* Not using CPAP for any reasons or patients on dental device but would like to try alternative treatments for OSA.
* Able to sign informed consent and use the PEEP nasal valve.
* Age between 18-65 years old.
* Willing to attend follow up.

Exclusion Criteria:

* Known nasal problems like deformities or significant rhinitis affecting application of PEEP nasal valve.
* Unable to sign consent or use PEEP nasal valve.
* Significant or unstable co-morbidities requiring other forms of treatment for OSA as priority.
* Coexisting sleep disordered breathing condition other than OSA requiring more complex treatment. E.g. central sleep apnea, significant Cheyne Stokes respiration or hypoventilation syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Apnea Hypopnea Index (AHI) | 1 month

SECONDARY OUTCOMES:
side effects as a measure of tolerability | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine and Therapeutics, Prince of Wales Hospital, CUHK, Shatin, Hong Kong